CLINICAL TRIAL: NCT00282750
Title: A Randomised Clinical Trial of a Bar-Coded Safety Sponge System
Brief Title: The Bar Coded Sponge Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Patient Safety Technologies, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2005-P-002344
Record Dates: First submitted 2006-01-26; First posted 2006-01-27 (Estimated); Last update posted 2010-01-14 (Estimated); Status verified 2010-01

CONDITIONS: Healthy
Keywords: "Surgery"[MeSH]; "Surgical Sponges"[MeSH]; "Automatic Data Processing"[MeSH]

INTERVENTIONS:
Device: Bar coded sponge and scanner

SUMMARY:
The purpose of this study is to test whether bar coded surgical sponges can significantly increase the safety of operations, specifically by (1) reducing discrepancies and miscounts, (2) reducing total staff time spent on sponge counting, and (3) reducing disruptions to the operating room as a system. Also, the study aims to further characterize the limitations of the current surgical sponge counting protocol.

DETAILED DESCRIPTION:
Prior work by Dr. Gawande showed that the incidence of a retained foreign body is between 1 in 9000 and 1 in 19000 inpatient operations, or at least once a year for a hospital of any size. Leaving foreign objects in body cavities after surgery can lead to infection, bowel obstruction and in some cases, death. The current approach to preventing this problem is based on adherence to a counting protocol to check the number of instruments and sponges at the beginning and end of the case. The problem of retained foreign body is often attributed to error in the counting process-for example in the case of a retained object, count totals at the beginning and end of the case can be erroneous if an item was not initially counted, or if an item was "double- counted" at the end of a case. In addition to this potential for incorrect counts, the counting protocols can lead to disruptions in case flow and inefficiencies.

In an observational study of surgical performance, which brought human factors experts into Brigham and Women's Hospital operating rooms to examine 10 complex cases, counting protocols for tracking instruments and sponges in particular played a surprisingly negative role on team performance. After the incision was made, nurses devoted an average of 35 minutes to the counting protocols. This represented 14.5% of the operative time. During this time, the investigators were able to document substantial negative effects on surgical work while the nurses were involved in the counting protocol. Furthermore, a counting discrepancy was observed to occur in two-thirds of the cases with a total of 17 discrepancies in 9 cases. As a result, in several patients, progress of a still-incomplete operation had to be substantially delayed or suspended while the nurses attempted to reconcile inconsistencies.

Based on these 2 studies, we conducted a rigorous search and innovation process, generating five possible technologies to detect when instruments or sponges are left behind. Discussions with engineers and a focus group of operating room nurses identified two of these technologies as most feasible for adoption: (1) bar-coded sponges; and (2) a computer vision system for tracking instruments.

SurgiCount Medical, which has subsequently joined Patient Safety Technologies, both of Los Angeles, has designed the Safety-sponge System, which utilizes bar-coded sponges and is now available for testing. The 4" x 4" X-ray detectable gauze sponges and 18" x 18" X-Ray detectable laparotomy pads are manufactured in the same fashion as sponges currently used today. They contain the X-ray detectable strip that can identify a retained sponge on a plain X-ray. A unique bar code (data matrix code) has been securely affixed to each sponge. The datamatrix code with ECC200 error correction allows for accuracy up to 1 error in 10.5 million (worst case), 1 in 612.9 million (best case). FDA 510K exemption status for the bar coded sponge has already been secured by the manufacturer. The bar code detector (sponge counter) has been designed as a small handheld computer with a touchscreen display.

Before introducing new technology into a healthcare system, it is important to study the effect that technology will have on the system. This includes both whether the new technology has the desired effect, but also whether there are any unintended negative effects. Our pre-clinical simulations suggest that the Safety-Sponge System has the potential to improve safety and efficiency in the operating room and other hospitals are moving ahead with purchase of the system. However we argue that the benefit must be proven in a randomized trial comparing it to the traditional counting protocol.

If our hypothesis is correct, this technology could revolutionize the counting procedures and improve both safety and efficiency in the operating room. This could decrease the risk of retained foreign bodies for patients. In addition, it could decrease the workload for the nursing staff in the operating room, leading to improvements in their working conditions and the overall safety of the system.

Comparisons: patients will be randomized to one of two equal groups: usual counting protocol versus bar-code technology assisted counting.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a scheduled general surgery (or subspecialty of general surgery) procedure in the general surgery operating room of the Brigham and Women's Hospital in Boston, MA, during the study period are eligible for enrollment in the study.
* Start times for eligible cases must be between 7AM and 3PM on a weekday.

Exclusion Criteria:

* Patients in the pre-op area who have already received pre-op sedation and have not yet been consented
* Patients who are undergoing a procedure by a specialty other than general surgery
* Patients whose procedure is being performed by a team whose members are not all trained to use the Bar Coded Sponge System
* After hours, weekend, add-on, or emergency cases
* Pregnant women
* Patients whose consent needs to be obtained through a surrogate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350
Dates: Start 2006-03; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
The amount of time per operating room staff member (circulating nurse and scrub technician) spent on sponge and instrument counts.
The phase of the counting episode (initial counts, objects added to field, closing counts, or repeat counts).
The number of and types of sponges added to the table during each counting event. Discrepancies, miscounts in the sponge count, and lost sponges during the course of the operation.
Time spent in search of a missing sponge or otherwise reconciling a counting discrepancy
A systems analysis of the O.R. during all counting procedures. Free-hand account of the counting procedure on a minute-to-minute basis which will include the following:
Team members present in the O.R. at the time of the time of the count and those actively involved in the counting procedure.
Concurrent activities in the O.R.
Any influence of the counting activity on the activities of other team members. These will include but are not limited to: (1) a request by the surgeon or other team member not being met, (2) a repeated request for assistance by another team member.
Any contributing factors. These will include but are not limited to: (1) original personnel not present in the O.R. due to a break or shift change, (2) conflict between team members, (3) communication breakdown.
The time of the entrance and exit of all team members from the room.
For intervention arm only, difficulties with the bar code technology or abandonment of the bar code technology will be recorded.
Request for an X-ray to rule out retained sponge will be noted, even if the X-ray is cancelled or not performed due to the risks of prolonged anesthesia time.
When an X-ray is requested, the following data points will be collected:
Time X-ray request made
Arrival time of X-ray technician in O.R.
Time X-ray results are available
When applicable, time X-ray request is cancelled and reason why

SECONDARY OUTCOMES:
Team survey at completion of case
To evaluate the ease and value of the Safety-Sponge System
To determine the confidence of the OR team in the Safety-Sponge System
To determine the team's evaluation of its own performance during the case. Specifically, whether the case went smoothly, whether there were any impediments to team performance, and if there was anyway that the team could have performed better.
Medical record review.
Medical record reviews will be performed to follow up on the patients' status sixty days after the surgical procedure. The presence or absence of retained sponges or instruments will be the measured outcome for chart review.

CONTACTS AND LOCATIONS:
Overall Officials: Atul A Gawande, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Gawande AA, Studdert DM, Orav EJ, Brennan TA, Zinner MJ. Risk factors for retained instruments and sponges after surgery. N Engl J Med. 2003 Jan 16;348(3):229-35. doi: 10.1056/NEJMsa021721. PMID 12529464
- [Background] Recommended practices for sponge, sharp, and instrument counts. AORN Recommended Practices Committee. Association of periOperative Registered Nurses. AORN J. 1999 Dec;70(6):1083-9. doi: 10.1016/s0001-2092(06)62224-2. No abstract available. PMID 10635432
- [Background] Christian CK, Gustafson ML, Roth EM, Sheridan TB, Gandhi TK, Dwyer K, Zinner MJ, Dierks MM. A prospective study of patient safety in the operating room. Surgery. 2006 Feb;139(2):159-73. doi: 10.1016/j.surg.2005.07.037. PMID 16455323